CLINICAL TRIAL: NCT01485133
Title: Water Colonoscopy Versus Air Colonoscopy for Unsedated Patients With Prior Abdominal or Pelvic Surgery: a Prospective Randomized, Controlled Trial
Brief Title: Water Method Colonoscopy in Patients With Prior Surgery
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: 20111103-9
Record Dates: First submitted 2011-11-30; First posted 2011-12-05 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Intubation; Surgery; Adenoma; Pain
Keywords: colonoscopy; water; surgery; unsedated
MeSH Terms: conditions — Adenoma; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Air colonoscopy: Colonoscopy will be performed without medications and with judicious air insufflation during colonoscope insertion.
- Water colonoscopy: Colonoscopy will be performed without medications and aided by water infusion in-lieu of air insufflation during insertion of the colonoscope. The water infusion involves putting warm sterile water into the colon to open up the colon for advancement of the colonoscope until the end of the colon (cecum) is reached. The water is delivered via a needle adaptor or the built-in scope irrigation channel by an infusion pump equipped with a foot switch which will be controlled by the endoscopist. Infused water used to cleanse residual fecal matter will be suctioned as needed to clear the colonic lumen.

SUMMARY:
Water method with water exchange has been shown to reduce medication requirement and pain experienced during colonoscopy. It increases the success rate of cecal intubation in sedated and unsedated patients undergoing screening colonoscopy. Exchange of water during scope insertion minimizes distension of the colonic lumen and decreases loop formation. Exclusion of air from the colon during insertion by omission of air insufflations and suction removal of residual air prevent elongation of the colon. These maneuvers facilitate colonoscopy insertion in average patients and may enhance the success of difficult colonoscopy.

Prior abdominal or pelvic surgery is an independent factor for difficult colonoscopy, the probable adhesion may change the anatomy and increase the discomfort of patients. We postulate that these patients may benefit from using the water method for colonoscopy. In this proposal we test the hypothesis that compared with conventional air insufflations the water method with water exchange significantly enhances the success rate of cecal intubation in patients with prior abdominal or pelvic surgery.

The aim of the study is to compare the outcome of colonoscopy using the water method versus the conventional air method in patients with prior abdominal or pelvic surgery. The primary outcome is cecal intubation success rate. The secondary outcomes include cecal intubation time, maximum pain score during colonoscopy, overall pain score after colonoscopy and adenoma detection rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prior abdominal or pelvic surgery,

Exclusion Criteria:

* History of colorectal surgery
* Severe colonic stricture or obstructing tumor
* Patients who cannot give informed consent and those who are hemodynamically unstable

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prior abdominal or pelvic surgery undergoing unsedated colonoscopy will be recruited in this study.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Cecal intubation success rate | up to ten months
  Insertion of a colonoscope to the cecum

SECONDARY OUTCOMES:
Adenoma detection rate | up to ten months
  The proportion of participants with at least one adenoma in each group
Pain Scores on the Visual Analog Scale | up to ten months
  0 = no pain, to 10 = most severe pain
Cecum intubation time | up to ten months
  Total time of colonoscope intubation from anus to cecum

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, MD, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Leung FW. Water exchange may be superior to water immersion for colonoscopy. Clin Gastroenterol Hepatol. 2011 Dec;9(12):1012-4. doi: 10.1016/j.cgh.2011.09.007. Epub 2011 Sep 22. No abstract available. PMID 21946120
- [Background] Leung FW, Leung JW, Mann SK, Friedland S, Ramirez FC. The water method significantly enhances patient-centered outcomes in sedated and unsedated colonoscopy. Endoscopy. 2011 Sep;43(9):816-21. doi: 10.1055/s-0030-1256407. Epub 2011 May 24. PMID 21611947
- [Background] Leung FW, Harker JO, Jackson G, Okamoto KE, Behbahani OM, Jamgotchian NJ, Aharonian HS, Guth PH, Mann SK, Leung JW. A proof-of-principle, prospective, randomized, controlled trial demonstrating improved outcomes in scheduled unsedated colonoscopy by the water method. Gastrointest Endosc. 2010 Oct;72(4):693-700. doi: 10.1016/j.gie.2010.05.020. Epub 2010 Jul 8. PMID 20619405
- [Background] Leung CW, Kaltenbach T, Soetikno R, Wu KK, Leung FW, Friedland S. Water immersion versus standard colonoscopy insertion technique: randomized trial shows promise for minimal sedation. Endoscopy. 2010 Jul;42(7):557-63. doi: 10.1055/s-0029-1244231. Epub 2010 Jun 30. PMID 20593332
- [Background] Leung JW, Mann SK, Siao-Salera R, Ransibrahmanakul K, Lim B, Cabrera H, Canete W, Barredo P, Gutierrez R, Leung FW. A randomized, controlled comparison of warm water infusion in lieu of air insufflation versus air insufflation for aiding colonoscopy insertion in sedated patients undergoing colorectal cancer screening and surveillance. Gastrointest Endosc. 2009 Sep;70(3):505-10. doi: 10.1016/j.gie.2008.12.253. Epub 2009 Jun 24. PMID 19555938
- [Derived] Luo H, Zhang L, Liu X, Leung FW, Liu Z, Wang X, Xue L, Wu K, Fan D, Pan Y, Guo X. Water exchange enhanced cecal intubation in potentially difficult colonoscopy. Unsedated patients with prior abdominal or pelvic surgery: a prospective, randomized, controlled trial. Gastrointest Endosc. 2013 May;77(5):767-73. doi: 10.1016/j.gie.2012.12.007. Epub 2013 Feb 5. PMID 23394837